CLINICAL TRIAL: NCT07022574
Title: Evaluating the Impact of Autoimmune Protocol Diet on Proteinuria in Patients With IgA Nephropathy
Brief Title: Autoimmune Protocol Diet Intervention on Proteinuria in IgA Nephropathy Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Thuy T. Tran, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 25-0145
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: IgA Nephropathy; Kidney disease; Low inflammation diet; Autoimmune Protocol Diet; Protein in urine; Autoimmune Kidney Disease; Elimination diet; Diet and Kidney disease
MeSH Terms: conditions — Glomerulonephritis, IGA; Kidney Diseases; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AIP Intervention arm (Experimental): Autoimmune Protocol Diet intervention
  Interventions: Behavioral: Low inflammation diet intervention

INTERVENTIONS:
Behavioral: Low inflammation diet intervention — Autoimmune Protocol Diet intervention
  Other Names: Autoimmune Protocol Diet

SUMMARY:
This study at UCLA Center for Health Sciences is testing whether the Autoimmune Protocol (AIP) diet can lower protein levels in the urine of people with IgA Nephropathy (IgAN), a common kidney disease that can lead to kidney failure. The AIP diet avoids foods that may cause inflammation (like dairy, grains, and sugar) for 8 weeks, then gradually reintroduces them over 4 months. We're enrolling 30 adults aged 18-65 with IgAN and protein in their urine to try this diet for 6 months. Participants will track their urine protein daily at home, keep a food log, and have monthly lab checkups, with support from a diet expert. The main goal is to see if the diet reduces urine protein by 20% or more, which could slow disease progression and reduce the need for treatments like dialysis. This exploratory study aims to find out if diet changes can help manage IgAN.

DETAILED DESCRIPTION:
This study, conducted at UCLA Center for Health Sciences, explores the potential of the Autoimmune Protocol (AIP) diet as a novel intervention for IgA Nephropathy (IgAN), a chronic kidney condition driven by immune system dysfunction. IgAN involves the deposition of galactose-deficient IgA1 (Gd-IgA1) in the glomeruli, triggering inflammation and progressive renal damage. Emerging evidence points to the gut, particularly the gastric-associated lymphoid tissue (GALT), as a key site where aberrant immune responses initiate this process. The AIP diet, a structured elimination and reintroduction plan, has shown promise in reducing inflammation in other autoimmune conditions like inflammatory bowel disease and rheumatoid arthritis. This study builds on a clinical observation of proteinuria reduction in an IgAN patient post-renal transplant following AIP diet adoption, aiming to test its broader applicability.

The intervention spans 6 months and is divided into two phases. The initial 8-week elimination phase removes foods known to provoke inflammation-such as dairy, grains, legumes, nightshades, and refined sugars-which may influence GALT activity and Gd-IgA1 production. This is followed by a 4-month reintroduction phase, where foods are systematically re-added to assess individual tolerances and their impact on renal markers. Unlike pharmacological approaches targeting downstream effects (e.g., ACE inhibitors) or upstream Gd-IgA1 production (e.g., Budesonide), the AIP diet offers a non-invasive strategy to modulate mucosal immunity. The study hypothesizes that reducing dietary inflammatory triggers could decrease immune complex formation, thereby lowering proteinuria and potentially altering disease trajectory.

Participants will receive extensive support, including initial training from a certified AIP nutritionist, two AIP cookbooks, and ongoing guidance via email or phone consultations. Daily home monitoring involves urine dipsticks to measure protein levels, complemented by weekly food journaling to track adherence and identify correlations with urinary changes. Monthly in-person visits will collect blood and urine samples for laboratory analysis, including Chem7, to assess renal function and metabolic health. This single-center, open-label design prioritizes feasibility and real-world applicability, with no placebo group, as the focus is on detecting a signal of efficacy in a small cohort.

The study's scientific foundation rests on the multi-hit pathogenesis model of IgAN, where mucosal immune dysregulation in the gut precedes renal injury. By targeting GALT, which constitutes a significant portion of the body's immune interface, the AIP diet may reduce the production of pathogenic IgA1. Previous dietary studies in IgAN, such as gluten-free interventions, have hinted at gut-renal connections, but none have tested a comprehensive low-inflammation approach like AIP. Technical considerations include the use of the urinary protein-to-creatinine ratio as a reliable, non-invasive marker of proteinuria, validated in nephrology research for its sensitivity to treatment effects.

Safety is a priority, with risks limited to mild discomfort from blood draws (e.g., bruising), dietary adjustment challenges, and minimal inconvenience from daily urine testing. Adverse events will be logged and reported per IRB standards, with monthly lab monitoring ensuring early detection of any renal or metabolic concerns. The study's exploratory nature and small sample size (n=30) aim to generate preliminary data, with statistical power calculated to detect a 20% proteinuria reduction.

Funded by individual donations, this research is independent of commercial interests, covering costs for lab tests, dietary education, and participant support materials. Findings will contribute to the growing understanding of diet's role in kidney disease management, with results shared through peer-reviewed journals and scientific conferences. This study represents a first step toward integrating dietary strategies into IgAN care, offering a low-risk, patient-centered complement to existing therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Diagnosed with IgA Nephropathy (IgAN)
* Active disease with urine protein/creatinine ratio ≥ 1
* Stable ARB or ACE inhibitor for at least 1 month prior
* GFR > 30
* Not on Budesonide 1 month prior or during study

Exclusion Criteria:

* Inability to comply with dietary or follow-up requirements
* Participation in other interventional studies
* Significant comorbidities interfering with study participation -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Urinary Protein to Creatine Ratio at 6months | 6 months
  Primary Outcome Measure
  1. Change in Urinary Protein-to-Creatinine Ratio
  * Description: This measure assesses the reduction in proteinuria, a key indicator of IgA Nephropathy (IgAN) activity, following the Autoimmune Protocol (AIP) diet intervention. The urinary protein-to-creatinine ratio (UPCR) will be calculated from spot urine samples collected at baseline and monthly intervals. The study aims to detect a reduction of 20% or greater from baseline, reflecting a clinically meaningful improvement in kidney function.
  * Time Frame: Baseline to 6 months (end of study).
  * Measurement: Expressed as grams of protein per gram of creatinine (g/g), analyzed via laboratory testing of urine samples.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD that underlie results in a publication.

REFERENCES:
- [Background] Konijeti GG, Kim N, Lewis JD, Groven S, Chandrasekaran A, Grandhe S, Diamant C, Singh E, Oliveira G, Wang X, Molparia B, Torkamani A. Efficacy of the Autoimmune Protocol Diet for Inflammatory Bowel Disease. Inflamm Bowel Dis. 2017 Nov;23(11):2054-2060. doi: 10.1097/MIB.0000000000001221. PMID 28858071